CLINICAL TRIAL: NCT00401180
Title: Phase I Trial of Weekly Docetaxel and Daily Temozolomide in Patients With Metastatic Disease
Brief Title: Docetaxel and Temozolomide in Treating Patients With Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert Bukowski, Cleveland Clinic Taussig Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-4737; P30CA043703 (NIH); CASE-CCF-4737
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2007-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Docetaxel; Temozolomide

INTERVENTIONS:
Drug: docetaxel — administered weekly in 5 escalating doses of 25 to 35 mg/ m(2) as a one-hour bolus intravenous infusion for 3 consecutive weeks.
Drug: temozolomide — administered orally daily for 3 weeks (escalating doses of 75 to 100 mg/m(2)). Cycles were repeated at 4 week intervals.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel and temozolomide in treating patients with metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity profile, dose-limiting toxicity, and maximum tolerated dose of docetaxel and temozolomide (TMZ) in patients with metastatic cancer.

Secondary

* Determine the activity of docetaxel and TMZ in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive docetaxel IV over 1 hour on days 1, 8, and 15 and oral temozolomide once daily on days 1-21. Treatment repeats every 28 days for up to 1 year in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of docetaxel and temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 6 patients receive treatment at the MTD.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of a nonhematologic malignancy that is refractory to standard therapy OR for which no standard therapy is available
* Measurable (by CT scan) or evaluable disease

  * If palliative radiotherapy has been administered, the measurable disease must be outside the radiation port
* Prior brain metastasis allowed provided it was definitely treated with external-beam radiotherapy, gamma knife, or surgical resection and is clinically stable

  * Repeat MRI or CT scans must demonstrate stabilization of disease 4 weeks after the definitive therapy is completed AND there must be no requirement for dexamethasone
* No active CNS metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 4 months
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL (epoetin alfa and/or transfusions allowed)
* Creatinine ≤ 2 mg/dL
* Bilirubin normal
* PT normal, unless the patient is on warfarin for prior deep vein thrombosis or pulmonary embolus, requiring INR maintained at 2.0 - 3.0
* Sodium and potassium normal
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* No decompensated cardiac arrhythmia or other severe cardiovascular disease (i.e., New York Heart Association [NYHA] class III-IV heart disease)

  * Patients with clinically stable NYHA class III or IV heart disease require cardiac clearance
* No peripheral neuropathy > grade 1
* No infection requiring IV antibiotics within the past 14 days
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No HIV positivity
* No hepatitis B surface antigen or hepatitis C antibody positivity
* No pulmonary embolus within the past 3 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 3 courses of prior immunotherapy and/or chemotherapy for metastatic disease

  * Interferon alfa in the adjuvant setting is not considered a course of prior therapy

    * Patients who relapse on adjuvant interferon alfa must be off therapy for ≥ 3 weeks
* No prior stem cell or organ transplantation
* More than 21 days since prior immunotherapy or chemotherapy
* At least 21 days since prior hormonal therapy (except luteinizing hormone-releasing hormone [LHRH] agonists) or radiotherapy and recovered
* More than 21 days since prior surgery requiring general anesthesia
* No concurrent radiotherapy
* Concurrent LHRH agonist therapy allowed
* Concurrent physiologic replacement steroids allowed
* No other concurrent chemotherapy or thalidomide
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF) during study chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 cycles
Dose-limiting toxicity | 4 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Bukowski, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Tamaskar I, Mekhail T, Dreicer R, Olencki T, Roman S, Elson P, Bukowski RM. Phase I trial of weekly docetaxel and daily temozolomide in patients with metastatic disease. Invest New Drugs. 2008 Dec;26(6):553-9. doi: 10.1007/s10637-008-9153-0. Epub 2008 Jul 15. PMID 18626572